CLINICAL TRIAL: NCT04434820
Title: External Negative Pressure Dressing System (ENPDS) vs. Traditional Wound Dressing for Cesarean Section Incision in Obese Women.
Brief Title: External Negative Pressure Dressing System vs. Traditional Wound Dressing for Cesarean Section Incision in Obese Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dalia Magdy Mokhtar, resident of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 642357
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Wound Dehiscence
Keywords: wound dehiscence; obesity; negative pressure therapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Basic information included age, ethnicity, weight, height, body mass index (BMI).
  Full obstetric, medical and surgical history. Informed written consent will be obtained Patients will receive standard preoperative antibiotic prophylaxis Wound dressing will be applied in a sterile fashion after primary closure of the Pfannenstiel incision closure by interrupted PROLENE Polypropylene Sutures The intervention group: placement of a sterile multilayer dressing (wicking fabric, reticulated foam, and occlusive adhesive). The dressing's tubing will then be attached to a (Yuwell 7E-A portable suction unit) that will deliver 125 mm Hg of continuous pressure to the dressing for 4 days.
  The comparison group: traditional sterile wound dressing of gauze and tape for 4 days.
  Post-operative data including: type of dressing used, postoperative hemoglobin, degree of pain, length of hospital stay, readmission for surgical site infection and the type of the surgical site infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- standard dressing group (No Intervention): patients will receive sterile wound dressing of gauze and tape for 4 days.
- External negative pressure dressing system group (Active Comparator): patients will receive placement of a sterile dressing of gauze and occlusive adhesive over the closed incision. The dressing's tubing will then be attached to a compact, portable negative-pressure therapy unit (Yuwell 7E-A portable suction unit) that will deliver -80 mm Hg of continuous pressure to the dressing and will remove exudates into a disposable canister for 4 days.
  Interventions: Device: External negative pressure dressing system (Yuwell 7E-A portable suction unit)

INTERVENTIONS:
Device: External negative pressure dressing system (Yuwell 7E-A portable suction unit) — A portable suction unit that will deliver 125 mm Hg of continuous pressure to the dressing and will remove exudates into a disposable canister for 4 days.
  Arms: External negative pressure dressing system group

SUMMARY:
Obesity is associated with increased cesarean section delivery rates and surgical site infections with associated increased post-operative morbidity, post-operative pain and length of hospital stay.

Negative pressure wound therapy (NPWT) technology could be used as a prophylactic measure to reduce surgical site infections in obese women undergoing cesarean section by immediate postoperative application in clean-contaminated, closed surgical incisions.

DETAILED DESCRIPTION:
Obesity, defined as body mass index (BMI, calculated as weight (kg)/ [height (m)] 2) of 30 or greater, is a common medical comorbidity of pregnancy affecting one third of reproductive-aged women. Maternal obesity is also a well-recognized risk factor for dysfunctional labor and cesarean delivery with a cesarean section rate of 33% in obese women with BMI of 30 or greater and 43% in women with BMIs of 40 or greater.

Obesity is an independent risk factor for post-operative surgical site infection. The risk of post-cesarean surgical site infection has been shown to double for every 5 unit increase in body mass index (BMI) above 30 kg/m , occurring in about 10% of obese women undergoing caesarean section despite prophylactic strategies (e.g. antibiotics).

This can be explained partly by a decreased blood flow in adipose tissue and an obesity-associated inflammation causing vascular dysfunction, which results in a local hypoxic response. Hypoxia impairs oxidative bacterial killing and leads to an increased risk of surgical site infection.

Wound healing is a sequence of physiologic events that include inflammation, epithelialization, fibroplasia, and maturation. Failure of wound healing at the surgical site can lead to seroma, hematoma, wound dehiscence, incisional hernia and surgical site infection.

Surgical site infection SSI according to The Centers for Disease Control and Prevention is as an infection occurring within 30 days from the operative procedure in the part of the body where the surgery took place, where there is purulent drainage from incision, isolated organisms from the incision, dehiscence or deliberate opening by the surgeon when the patient has at least one sign or symptom of clinical infection: localized pain, edema, erythema, warmth and fever greater than 38 c (unless culture of incision is negative) or there is an abscess or other evidence of infection is found during examination of incision, reoperation, or pathologic or radiologic exam.

SSIs is divided into incisional SSI and organ/space SSI. Incisional SSI is further divided into superficial and deep incisional SSI. Superficial Incisional Surgical Site Infection involves skin or subcutaneous tissue cellulitis, seroma, hematoma, wound healing disruption, or dehiscence. Deep Incisional Surgical Site Infection involves deep soft tissues such as fascia or muscle within incision. Organ/Space Surgical Site Infection involves any part of the anatomy other than the incision. SSI is associated with a maternal mortality rate of up to 3%.

Wound complication, even if not accompanied by an infection, is a significant cause of postoperative morbidity following cesarean delivery. In addition to the increased cost of care, there is the inconvenience of therapy, increased postoperative pain and convalescence, as well as difficulty with activities of daily living.

It is logical to employ novel risk reducing approaches including negative pressure wound therapy at the time of surgery that may prevent wound complications and to ensure that there is a demonstrable benefit to their use for wound complication prophylaxis.

Negative pressure wound therapy (NPWT), also known as a vacuum assisted closure (VAC), involves the controlled application of sub-atmospheric pressure to the local wound environment, using a sealed wound dressing connected to a vacuum to promote healing by primary intention by reducing the risk of hematoma / seroma due to improved lymphatic drainage and reduces the risk of wound dehiscence by decreasing the lateral and shear stress on sutures and decreasing bacterial load and wound fluids and by increasing blood flow, oxygenation, angiogenesis, and epithelialization.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 or older
* BMI: 30 or greater
* undergoing Cesarean section through a Pfannenstiel incision

Exclusion Criteria:

* Prolonged Rupture of membranes >18 hours
* Intra amniotic infection
* Severe anemia
* Vasculopathies as in hypertension/pre-eclampsia, pregestational / gestational diabetes mellitus, smoking and substance abuse
* Prolonged steroids therapy as in SLE, ITP
* Intraoperative complications as bladder or bowel injury , placenta previa / accreta, difficult fetal extraction , ovarian cysts, pelvic abscess
* Intra-abdominal or subcutaneous drain

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 260 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
incidence of wound dehiscence | till 30 days post operative
  separation of the incision line prior to complete healing resulting in an open wound.

SECONDARY OUTCOMES:
post operative pain | till 30 days post operative
  post-operative pain assessed by Wong-Baker Faces pain rating scale,from 0=no pain to 10=maximal pain
length of hospital stay | till 30 days post operative
  days spent admitted to the hospital
the need for re-admission | till 30 days post operative
  if the patient encountered surgical site infection requiring re admission to the hospital
further need for additional antibiotics | till 30 days post operative
  if the surgical site infection required additional post operative antibiotics
peri-incision blistering | till 30 days post operative
  if any skin blistering occurs under the occlusive adhesive layer
patient mobility | 4 days
  if attachment to a negative pressure pump affects patients mobility
surgical site infection | 30 days post operative
  as defined by the CDC

CONTACTS AND LOCATIONS:
Overall Officials: Dalia M Mokhtar, MBBCh, Principal Investigator — resident of obstetrics and gynecology; Marwan O Elkady, MD, Study Director — Lecturer of obstetrics and gynecology; Mohammed S El Sokkary, MD, Study Chair — Professor of obstetrics and gynecology
Locations (1):
- AinShams maternity hospital, Cairo, Al-Waili, Egypt

IPD SHARING:
Plan to Share IPD: Yes
patient's age ,ethnicity,gravidity,parity,gestational age ,previous cesarean section, previous surgeries,weight, height,BMI,pre/post operative haemoglobin,degree of post operative pain,incidence and type of surgical site infection,length of hospital stay, need for re-admission,need for additional antibiotics
Supporting Information: Study Protocol, SAP
Time Frame: after completing the study and henceforth .
Access Criteria: everyone can review the IPD on this site for any type of analysis they desire .

REFERENCES:
- [Background] Hyldig N, Vinter CA, Kruse M, Mogensen O, Bille C, Sorensen JA, Lamont RF, Wu C, Heidemann LN, Ibsen MH, Laursen JB, Ovesen PG, Rorbye C, Tanvig M, Joergensen JS. Prophylactic incisional negative pressure wound therapy reduces the risk of surgical site infection after caesarean section in obese women: a pragmatic randomised clinical trial. BJOG. 2019 Apr;126(5):628-635. doi: 10.1111/1471-0528.15413. Epub 2018 Sep 7. PMID 30066454
- [Background] Mark KS, Alger L, Terplan M. Incisional negative pressure therapy to prevent wound complications following cesarean section in morbidly obese women: a pilot study. Surg Innov. 2014 Aug;21(4):345-9. doi: 10.1177/1553350613503736. Epub 2013 Sep 20. PMID 24056202
- [Background] Orth TA, Gerkovich MM, Heitmann E, Overcash J, Gibbs C, Parrish M. Cesarean Delivery with External Negative Pressure Dressing System: A Retrospective Cohort Study. Surg J (N Y). 2016 Jul 20;2(3):e59-e65. doi: 10.1055/s-0036-1585470. eCollection 2016 Jul. PMID 28824992
- [Background] Scalise A, Tartaglione C, Bolletta E, Calamita R, Nicoletti G, Pierangeli M, Grassetti L, Di Benedetto G. The enhanced healing of a high-risk, clean, sutured surgical incision by prophylactic negative pressure wound therapy as delivered by Prevena Customizable: cosmetic and therapeutic results. Int Wound J. 2015 Apr;12(2):218-23. doi: 10.1111/iwj.12370. Epub 2014 Sep 19. PMID 25234139
- [Background] Smid MC, Dotters-Katz SK, Grace M, Wright ST, Villers MS, Hardy-Fairbanks A, Stamilio DM. Prophylactic Negative Pressure Wound Therapy for Obese Women After Cesarean Delivery: A Systematic Review and Meta-analysis. Obstet Gynecol. 2017 Nov;130(5):969-978. doi: 10.1097/AOG.0000000000002259. PMID 29016508
- [Background] Todd B. New CDC Guideline for the Prevention of Surgical Site Infection. Am J Nurs. 2017 Aug;117(8):17. doi: 10.1097/01.NAJ.0000521963.77728.c0. PMID 28749874
- [Background] Wells CI, Ratnayake CBB, Perrin J, Pandanaboyana S. Prophylactic Negative Pressure Wound Therapy in Closed Abdominal Incisions: A Meta-analysis of Randomised Controlled Trials. World J Surg. 2019 Nov;43(11):2779-2788. doi: 10.1007/s00268-019-05116-6. PMID 31396673
- [Background] Zuarez-Easton S, Zafran N, Garmi G, Salim R. Postcesarean wound infection: prevalence, impact, prevention, and management challenges. Int J Womens Health. 2017 Feb 17;9:81-88. doi: 10.2147/IJWH.S98876. eCollection 2017. PMID 28255256